CLINICAL TRIAL: NCT03725293
Title: Randomized Comparative Evaluation of Midline Catheters for Thrombophlebitis
Brief Title: Midlines and Thrombophlebitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Principal Investigator, Amit Bahl, Director, Emergency Ultrasound, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-379
Record Dates: First submitted 2018-10-25; First posted 2018-10-31 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Catheter Infection; Catheter Thrombosis; Catheter Complications
Keywords: thrombosis; superficial venous thrombosis; deep venous thrombosis; line related infection; catheter survival
MeSH Terms: conditions — Thrombosis; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Prospective single-site, parallel, two-arm, randomized investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Angiodynamics BioFlo Midline Catheter (Active Comparator): Placement of clinically indicated Angiodynamics BioFlo midline catheter.
  Interventions: Device: Angiodynamics BioFlo Midline Catheter
- Teleflex Arrowg+ard Blue Advanced Midline Catheter (Active Comparator): Placement of clinically indicated Teleflex Arrowg+ard Blue Advanced Midline Catheter
  Interventions: Device: Teleflex Arrowg+ard Blue Advanced Midline Catheter

INTERVENTIONS:
Device: Angiodynamics BioFlo Midline Catheter — Placement of Angiodynamics BioFlo Midline Catheter.
  Arms: Angiodynamics BioFlo Midline Catheter
Device: Teleflex Arrowg+ard Blue Advanced Midline Catheter — Placement of Teleflex Arrowg+ard Blue Advanced Midline Catheter.
  Arms: Teleflex Arrowg+ard Blue Advanced Midline Catheter

SUMMARY:
Peripherally inserted central catheters (PICCs) are central catheters that are placed via peripheral vein under ultrasound guidance and may be used for patients with difficult venous access for long-term central or peripheral infusion therapies as well as central venous pressure monitoring in a critical care setting. Although PICCs provide a great option for some patients, these catheters have known complications including catheter-related bloodstream infection, catheter-related venous thrombosis or clotting, malfunction, and high cost. Midline catheters represent a potentially attractive alternative to PICCs for peripheral infusions. As midlines have increased in popularity and new midlines have been introduced into the market, it is necessary to better understand complication profiles of various midline catheters, as it is likely that all catheters are not created equal. Specifically, the incidence of symptomatic catheter-related thrombosis is of interest. Some midline catheters are coated to provide protection against catheter-related venous thrombosis and/or catheter-related bloodstream infection. The theoretical benefit(s) of these catheters need further validation in human subjects.

DETAILED DESCRIPTION:
Study Design

The investigators propose a prospective single-site, parallel, two-arm, randomized investigation to assess catheter-related symptomatic upper extremity venous thrombosis (CR-UEVT), catheter-related bloodstream infection, and functionality of two single lumen midline catheters: AngioDynamics BioFlo 4 F and Teleflex Arrowg+ard Blue Advance 4.5 F.

Research staff of Beaumont Health Institute will allocate two midline catheters to eligible participants according to a pre-generated randomized list at a 1:1 ratio in block randomization to AngioDynamics BioFlo or Tele-flex Arrowg+ard Blue Advanced midline catheters. Participant enrollment will take place from November 2018 until recruitment of 250 participants, 125 in each group, is complete. Demographic and health-related information will be obtained from electronic medical records during enrolled period at William Beaumont Hospital.

Practitioner Participation/Training

Advanced Practice Providers within the bedside PICC/Midline service at the Royal Oak campus are eligible to place catheters for this study. All investigators are credentialed in placing PICCs and midlines by institutional policy and have greater than one year of experience in these procedures.

Initial Assessment

Post-cannulation and post securement, functionality is confirmed with blood sampling (10 cc) and flush without resistance.

The research team also will document practitioner details, the vascular access device (VAD) used, the time of VAD placement, number of attempts, need for a rescue inserter, the vein that was cannulated, depth and diameter of the vein, and the indication for VAD placement. An attempt is defined as each time the needle punctures the skin. Data will be collected from the electronic medical record and includes: age, gender, body mass index (BMI), vital signs, relevant past medical history. Indication for catheter placement will also be recorded.

Follow-up Assessment

Investigators will perform a follow-up assessment on all catheters within 24 hours of insertion and then daily for the life of the VAD. At each follow-up interval, the researcher will document the time of evaluation and assessment of functionality as well as review the patient chart for signs and symptoms of catheter-related bloodstream infection. If the catheter was identified to have failed during follow-up assessment the date and time of failure and the reason for failure will be documented. For all failed catheters, re-insertion attempt data will be tracked through the medical record.

Superficial venous thrombosis (SVT) and deep venous thrombosis (DVT) rates will be calculated based on upper extremity proven diagnosis of SVT and/or DVT in symptomatic cases. Radiology interpretations will be reviewed for findings consistent with CR-UEVT.

Infection rate will be tracked using confirmed catheter-related blood stream infection data from the surveillance team within the epidemiology department. The team utilizes the CDC definition of laboratory-confirmed blood-stream infection (LCBSI).

The medication administration record will be queried for all medications given through each catheter.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients 18 years of age and older
* Inpatients that require midline catheter placement by the bedside vascular access team

Exclusion Criteria:

* Do not meet inclusion criteria
* Multiple lumens required
* Alternative diameter of catheter used
* If already enrolled once prior
* Withdraw voluntarily from the study
* Actively (within 24 hours) taking a therapeutic dose of an anticoagulant (heparin, low molecular weight heparin, enoxaparin, rivaroxaban, apixaban, dabigatran, edoxaban, warfarin, arixtra, factor Xa inhibitors)
* Receiving a midline catheter for anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bahl, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Hospital - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahl A, Johnson S, Mielke N, Chen NW. Risk Factors for Coated Midline Catheter-Related Thrombosis: A Secondary Analysis of Existing Trial Data. J Infus Nurs. 2023 Sep-Oct 01;46(5):259-265. doi: 10.1097/NAN.0000000000000518. PMID 37611283
- [Derived] Bahl A, Diloreto E, Jankowski D, Hijazi M, Chen NW. Comparison of 2 Midline Catheter Devices With Differing Antithrombogenic Mechanisms for Catheter-Related Thrombosis: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2127836. doi: 10.1001/jamanetworkopen.2021.27836. PMID 34613402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Angiodynamics BioFlo Midline Catheter | Teleflex Arrowg+Ard Blue Advanced Midline Catheter
Started | 106 | 106
Completed | 94 | 97
Not Completed | 12 | 9
Not completed — Physician Decision | 9 | 6
Not completed — alternative vascular access needs | 1 | 2
Not completed — venous anatomy screen failures | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Angiodynamics BioFlo Midline Catheter | Teleflex Arrowg+Ard Blue Advanced Midline Catheter | Total
Number analyzed (Participants) | 94 | 97 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.29 (16.3) | 59.5 (17.1) | 60.2 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 40 | 37 | 77
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94 | 97 | 191

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity CR-UEVT
Description: Number of participants with proven sonographic diagnosis of DVT and/or SVT
Time Frame: 30 days post line insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Angiodynamics BioFlo Midline Catheter | Teleflex Arrowg+Ard Blue Advanced Midline Catheter
Number analyzed (Participants) | 94 | 97
Participants | 7 | 11

2. Secondary Outcome: Line Related Infection
Description: Number of participants with catheter related laboratory confirmed bloodstream infection per Centers for Disease Control (CDC) guidelines
Time Frame: 30 days post line insertion
Measure: Count of Participants; unit: Participants
Arm/Group | Angiodynamics BioFlo Midline Catheter | Teleflex Arrowg+Ard Blue Advanced Midline Catheter
Number analyzed (Participants) | 94 | 97
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days post line insertion
Arm/Group | Angiodynamics BioFlo Midline Catheter | Teleflex Arrowg+Ard Blue Advanced Midline Catheter
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/97
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/97
Other Adverse Events (participants affected / at risk) | 22/94 | 20/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiodynamics BioFlo Midline Catheter (N=94) | Teleflex Arrowg+Ard Blue Advanced Midline Catheter (N=97)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Angiodynamics BioFlo Midline Catheter (N=94) | Teleflex Arrowg+Ard Blue Advanced Midline Catheter (N=97)
Catheter Failure (Blood and lymphatic system disorders) | 22 | 20 — Catheter failure prior to completion of therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03725293/Prot_SAP_000.pdf